CLINICAL TRIAL: NCT01415414
Title: The Image Quality and Radiation Dose of CECT With Ultravist® in Patients With Abdominal Pelvic Disease - INDEX
Brief Title: Observational Study of Ultravist in Patients Requiring CECT
Acronym: INDEX
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15515; UV1011CN (Other: Company Internal)
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Diagnostic Imaging
Keywords: Image quality; CNR; SNR; Abdominal; Pelvic
MeSH Terms: interventions — iopromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)

INTERVENTIONS:
Drug: Iopromide (Ultravist, BAY86-4877) — CT enhancement for abdominal or pelvic scan. Generally doses of up to 1.5 g iodine per kg body weight are well tolerated

SUMMARY:
It is a prospective, non-interventional, multi-center study. The primary objective of this study is to evaluate the image quality of Ultravist in patients requiring contrast-enhanced CT considering the routine use in patient population's, region's indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing contrast enhanced CT Imaging with Ultravist (iopromide) in abdomen or pelvis.

Exclusion Criteria:

* There is no other exclusion criteria beyond the contraindications contained in the Summary of Product Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing contrast enhanced CT Imaging with Ultravist (iopromide) in abdomen and pelvis, including relevant vessels
Sampling Method: Probability Sample
Enrollment: 11660 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Image quality evaluated by calculated CNR (Contrast to Noise Ratio) | 1 day

SECONDARY OUTCOMES:
Image quality evaluated by calculated SNR (Signal Noise Ratio) | 1 day
Descriptive analysis of contrast medial injection protocol | 1 day
Radiation dose (CTDIvol) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China